CLINICAL TRIAL: NCT06056674
Title: Unified Protocol for Preventing Emotional and Academic Challenges in Education (U-PEACE) Randomized Controlled Trial
Brief Title: Unified Protocol for Preventing Emotional and Academic Challenges in Education (U-PEACE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Institute of Educational Sciences (IES) (Unknown)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20230796
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Emotions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- U-PEACE Group (Experimental): Participants in this group will receive the U-PEACE intervention (study participation to last approximately 13 weeks).
  Interventions: Behavioral: U-PEACE Intervention
- Services As Usual (SAU) Group (Active Comparator): Participants in this group will receive service as usual (study participation to last approximately 13 weeks).
  Interventions: Behavioral: SAU

INTERVENTIONS:
Behavioral: U-PEACE Intervention — This program will involve about 13 group sessions, with each group session lasting approximately 40-50 minutes. The program session will be held about 2 times a week during the school day (e.g., lunch time) if the group meets in person, or at a pre-scheduled time every week if the group meets online via Zoom.
  Participants will learn how to better understand emotional experiences and use this understanding to embrace agency in challenging situations. Participants will develop skills to better deal with emotions by increasing awareness of what is happening in different settings and choose how to respond. Skill-building exercises may include mindfulness practices, flexible thinking, behavioral activation, problem-solving, and exposure activities.
  Arms: U-PEACE Group
Behavioral: SAU — Participants in this group will continue to receive standard of care within their school clinic.
  Arms: Services As Usual (SAU) Group

SUMMARY:
The purpose of the study is to evaluate the feasibility and effectiveness of a program for high school students with emotional and academic challenges U-PEACE and gaining feedback on that program.

ELIGIBILITY:
Inclusion Criteria:

Youth:

1. Adolescents between the ages of 13 and 18 years at the time of enrollment, who:

   1. display depressive symptoms above the clinical cut-off of 9 or above on the Patient Health Questionnaire-8 (PHQ-8),
   2. display elevated anxiety symptoms of 10 or above on the Generalized Anxiety Disorder 7-item Scale (GAD-7; Spitzer et al., 2006),
   3. are enrolled at the target High Schools (HS),
   4. have expressed interest in participating in the study, and
   5. have a caregiver who is available to sign study consent forms (if under 18 years of age)
2. Adolescents must be, or are willing to be, consented to receive services through School Health Initiative (SHI) (i.e., SHI consent). If they are under 18 years of age, their caregiver must provide consent.
3. Adolescents and caregivers are able to complete all study procedures in English or Spanish.

Teachers:

1. Individuals who are 18 years or older.
2. Individuals who are currently employed at the target HSs.
3. Individuals who are able to speak, read, and understand English.

Youth Exclusion Criteria:

1. The following individuals may be excluded at any time (e.g., before consent, after being enrolled).

   1. Individuals who do not wish to participate in this study and/or who are not able to read and understand the consent/assent.
   2. Individuals with self- or caregiver-reported history of seizures, neurological problems, autism spectrum disorder, substance use disorder, or serious mental illness (e.g., schizophrenia), and any indicator of a significant cognitive delay that would make U-PEACE inappropriate (e.g., full-time special education placement)
   3. Individuals with current anxiety or depressive symptoms or active suicidality at levels where more intensive services (e.g., day treatment, inpatient) would be warranted (e.g., hospitalization for suicidal behavior in the last 12 months).
2. Ineligible adolescents will be provided referrals to medical providers at the SHI, community agencies contracted with the Miami-Dade County Public Schools (M-DCPS) Office of Mental Health Services or emergency room settings, as appropriate.
3. Unclear cases will be reviewed by the PI and Director of the SHI, Co-I Lisa Gwynn, D.O.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Adolescent Academic Problems Checklist (AAPC) | At baseline, mid (approximately week 4), post (approximately week 9) and 1-month follow-up (approximately week 13)
  Scores on each item range from 0 to 3, with higher scores indicating more academic problems.
Therapeutic Alliance Scale for Children, Revised (TASC-R) | Mid (approximately week 4)
  Scores on each item range from 1 (not true) to 4 (very much true). This scale measures the perceived therapeutic alliance between child and therapist.
Client Satisfaction Questionnaire (CSQ) | Mid (approximately week 4)
  Total Scores range from 8 to 32, with higher scores indicating greater client satisfaction. The CSQ support used to evaluate satisfaction with a particular intervention, client self-efficacy and the likelihood of recommending the intervention to others.
Top Problems Assessment - Child Report as measured by Likert Scale | Up to 13 weeks
  The Top Problems assessment is used to identify self-reported target problems for treatment and track changes in problem severity over time. Identified top problem statements are rated on Likert scale from 0 (not at all a problem) to 10 (a huge problem).
Adherence to U-PEACE, as Measured by Homework Completion | At all group sessions (up to 9 weeks)
  Adherence to U-PEACE will be measured by the overall number of homework assignments completed.
Adherence to U-PEACE, as Measured by Session Attendance | At all group sessions (up to 9 weeks)
  Adherence to U-PEACE will be measured by the overall number of sessions attended.
Change in Revised Children's Anxiety and Depression Scale - Child Revised Short Version (RCADS-C-S) | At baseline, mid (approximately week 4), post (approximately week 9) and 1-month follow-up (approximately week 13)
  The Change in Revised Children's Anxiety and Depression Scale - Child Revised Short Version (RCADS-25) is 25-item self-reported scale measuring symptoms of anxiety and depression in youth. Items are rated on a 4-point scale from 1 (Never) to 4 (always) with total composite scores ranging from 0 to 75. A score of 70 or higher indicates high severity.
Change in Generalized Anxiety Disorder 7-item Scale (GAD-7) | At baseline, mid (approximately week 4), post (approximately week 9) and 1-month follow-up (approximately week 13)
  GAD-7 evaluates core anxiety concerns across a 7-item self-report measure. Items are rated using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). It yields a total score and a rating of impairment
Change in Patient Health Questionnaire 9-item Scale (Modified for Major Depressive Disorder in Adolescents; PHQ-9M) | At baseline, mid (approximately week 4), post (approximately week 9) and 1-month follow-up (approximately week 13)
  PHQ-9 evaluates core depression symptoms across 9 items. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day)

SECONDARY OUTCOMES:
School Achievement, as measured by attendance | Up to approximately 13 weeks
  Attendance is defined as number of days attending school (not absent)
School Achievement, as measured by report card | Up to approximately 13 weeks
  School achievement will be measured by a numeric score on each participant's school report card
Change in Child Anxiety Impact Scale-Academic Subscale (CAIS-AS) | At baseline, mid (approximately week 4), post (approximately week 9) and 1-month follow-up (approximately week 13)
  CAIS-AS is a youth- and caregiver-report measure that assesses the impact of anxiety on function. The Academic sub scale assesses the impact of anxiety on assignments and tests, getting to school on time, etc. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (very much), with higher scores indicating greater impact of anxiety symptoms on academics
Change in Affective Reactivity Scale (ARI) | At baseline, mid (approximately week 4), post (approximately week 9) and 1-month follow-up (approximately week 13)
  ARI is a 7-item youth- and caregiver-report measure of irritability. Items are rated on a 3-point Likert scale from 0 (not true) to 2 (certainly true)
Change in Distress Tolerance Scale (DTS) | At baseline, mid (approximately week 4), post (approximately week 9) and 1-month follow-up (approximately week 13)
  DTS is a 15-item youth report measure to evaluate emotional distress tolerance. Items are rated on a 5-point Likert scale from 1 (strongly agree) to 5 (strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Velez CV, Campez-Pardo M, Canovas JM, Pedronzo PM, Ahn YA, Dale CF, Dale SK, Gwynn L, Jensen-Doss A, Pulgaron ER, St George SM, Ehrenreich-May J. An Iteratively Adapted Transdiagnostic Prevention Program for Diverse High School Settings (U-PEACE): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 24;14:e74080. doi: 10.2196/74080. PMID 40990367